CLINICAL TRIAL: NCT05159544
Title: A Prospective, Multicenter, Noninterventional Cohort Study of Muti-Omics Models for Pan-Cancer Screening
Brief Title: The FuSion Program: A Prospective and Multicenter Cohort Study of Pan-Cancer Screening in Chinese Population
Status: Recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: FuSion
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: Muti-omics; Pan-cancer screening; Early detection
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Multi-omics model developing and training arm: Blood samples and individual health information from 50,000 participants in community, who got 3-year follow-up are selected.
- Multi-omics model validating arm: 10,000 participants in routine annual physicals from hospitals will be selected, and they will be followed up for 2 years.
- Multi-omics model evaluating arm: Participants in Taizhou cohort will be selected.

SUMMARY:
The integrative study by Fudan and Singlera for cancer early detection(The FuSion Program ) will evaluate sensitivity,specificity and positive/negative predictive value of the screening model jointly developed by FuDan University and Singlera in a 2-year follow-up corhort including 10,000 persons in routine annual physicals from dozens of hospitals. The multi-omics model for pan-cancer screening will be developed in a 3-year follow-up corhort including 50,000 natural persons in community containing genetic information of tumor families, assessment of epidemiological risk factors, tumor markers, proteomics, genomics and DNA methylation. After optimizing, the ability of this model will be validated in the Taizhou corhort in reality.

ELIGIBILITY:
Inclusion Criteria:

1. Take physical examinations in our research centers and have no cancer history;
2. "Population Health tracking Survey - simplified version of the questionnaire" must be filled according to the research program and an annual physical examination can be received as follow-up ;
3. Timely feed back the information related to tumor diagnosis in other hospitals to the investigator during the program;
4. Have no birth plan for the last 3 years;
5. Fully understand the study and voluntarily sign the informed consent.

Exclusion Criteria:

1. Have been diagnosed with esophageal cancer, gastric cancer, colorectal cancer, liver cancer, lung cancer, pancreatic cancer, breast cancer (including non-primary, such as recurrence, metastasis or other complications) and other malignant tumors;
2. Received blood transfusion, transplantation and other major operations within 3 months;
3. Participated in other interventional clinical researchs within 3 months;
4. Pregnant or lactating women;
5. Patients with autoimmune diseases, genetic diseases, mental diseases/disabilities and other diseases considered unsuitable for the study by the investigator;
6. Due to poor compliance, the researcher judged that the study could not be completed.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the communities in Taizhou city and medical centers in different provinces, including normal healthy people, high-risk people, those with benign disease and malignant diseases.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-07-06 (Estimated); Study Completion 2024-12-07 (Estimated)

PRIMARY OUTCOMES:
To develop a multi-omics model for pan-cancer screening integrating the markers of ctDNA mutation, DNA fragmentation and methylation et al. | assessed up to 36 months
  To construct a multi-dimensional ensembled stacked machine learning approach, employing several different base models on ctDNA mutation, DNA fragmentation and mehylation, to provide an effective model for cancer early detection.
To evaluate sensitivity,specificity,positive/negative predictive value of the screening model in participants taking routine annual physicals | assessed up to 24 months
  Sensitivity: the ability of a test to correctly identify patients with a disease. Specificity: the ability of a test to correctly identify people without the disease. Positive predictive value refers to the probability of the person having the disease when the test is positive. Negative predictive value refers to the probability of the person not having the disease when the test is negative.
To validate model's efficacy and clinical value in the diagnosis of cancers in Taizhou cohort. | assessed up to 12 months
  Cancer early detection could increase detection of cancer at early stages, when survival outcomes are better and treatment costs are lower. we will explore whether this model with high specificity could potentially improve long-term health outcomes and reduce cancer treatment costs.

CONTACTS AND LOCATIONS:
Overall Officials: Xingdong Chen, Ph.D, Study Director — Fudan University Taizhou Institute of Health Sciences, Taizhou, China; Rui Liu, Ph.D, Principal Investigator — Singlera Genomics Inc.
Locations (12):
- China (12):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Union Hospital affiliated to Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Taizhou Institute of Health Sciences, Taizhou, China, Taihou, Jiangsu
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Gole J, Gore A, He Q, Lu M, Min J, Yuan Z, Yang X, Jiang Y, Zhang T, Suo C, Li X, Cheng L, Zhang Z, Niu H, Li Z, Xie Z, Shi H, Zhang X, Fan M, Wang X, Yang Y, Dang J, McConnell C, Zhang J, Wang J, Yu S, Ye W, Gao Y, Zhang K, Liu R, Jin L. Non-invasive early detection of cancer four years before conventional diagnosis using a blood test. Nat Commun. 2020 Jul 21;11(1):3475. doi: 10.1038/s41467-020-17316-z. PMID 32694610